CLINICAL TRIAL: NCT00879996
Title: A Randomized Controlled Trial Comparing Buprenorphine and Methadone for Opioid Dependent Chronic Pain Patients
Brief Title: Buprenorphine and Methadone for Opioid Dependent Chronic Pain Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Richard Blondell, MD, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMD0350908A; K23AA015616 (NIH); R03DA029768 (NIH)
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Results first posted 2012-07-09 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Opiate Addiction
Keywords: Opiate Addiction; Narcotic Addiction; Drug Addiction; Pain
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders; Substance-Related Disorders; Pain | interventions — Methadone; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Methadone 10-60 mg per day in 2-4 divided doses for 6 months
  Interventions: Drug: Methadone
- 2 (Experimental): Buprenorphine 4-16 mg per day in 2-4 divided doses for 6 months (using tablets of buprenorphine/naloxone:4/1 mg)
  Interventions: Drug: Buprenorphine/naloxone

INTERVENTIONS:
Drug: Methadone — Oral, 10-60 mg per day, 2-4 times per day, 6 months
  Other Names: Dolophine
  Arms: 1
Drug: Buprenorphine/naloxone — Sub-lingual, 4-16 mg per day, divided 2-4 times/day, 6 months
  Other Names: Suboxone
  Arms: 2

SUMMARY:
The purpose of this study is to determine if buprenorphine or methadone is better for the treatment of chronic pain among patients who have become addicted to prescription narcotics.

DETAILED DESCRIPTION:
The purpose of this randomized clinical trial is to compare methadone with buprenorphine for the treatment of chronic pain among patients who have developed a physical dependence on prescription opiate analgesics that is associated with psychosocial dysfunction (i.e., addiction).

ELIGIBILITY:
Inclusion Criteria:

* chronic back pain
* opioid addiction
* not successful with abstinence
* at least 18 years old
* able to understand spoken English
* live in Western New York State (Erie or Niagara county)
* have health insurance or ability to pay for health care
* no methadone or buprenorphine treatment within past year
* not member of a vulnerable population (e.g., pregnancy, prisoner)

Exclusion Criteria:

* homelessness
* unable to give consent (e.g., dementia, psychosis)
* serious heart or lung disease
* taking a medication that could interact with methadone or buprenorphine
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Blondell, MD, Principal Investigator — SUNY Buffalo
Locations (2):
- United States (2):
  - Sheehan Memorial Hospital, Buffalo, New York
  - Erie County Medical Center, Buffalo, New York

REFERENCES:
- [Derived] Nielsen S, Tse WC, Larance B. Opioid agonist treatment for people who are dependent on pharmaceutical opioids. Cochrane Database Syst Rev. 2022 Sep 5;9(9):CD011117. doi: 10.1002/14651858.CD011117.pub3. PMID 36063082
- [Derived] Neumann AM, Blondell RD, Jaanimagi U, Giambrone AK, Homish GG, Lozano JR, Kowalik U, Azadfard M. A preliminary study comparing methadone and buprenorphine in patients with chronic pain and coexistent opioid addiction. J Addict Dis. 2013;32(1):68-78. doi: 10.1080/10550887.2012.759872. PMID 23480249

RESULTS

PARTICIPANT FLOW:
Groups:
- Methadone: Methadone 10-60 mg per day in 2-4 divided doses for 6 months
- Buprenorphine/Naloxone: Buprenorphine 4-16 mg per day in 2-4 divided doses for 6 months (using tablets of buprenorphine/naloxone:4/1 mg)
Period: Overall Study
Arm/Group | Methadone | Buprenorphine/Naloxone
Started | 28 | 26
Completed | 13 | 13
Not Completed | 15 | 13
Not completed — Lost to Follow-up | 7 | 6
Not completed — non-compliance | 6 | 4
Not completed — Physician Decision | 1 | 2
Not completed — psychiatric problem | 0 | 1
Not completed — put on parole | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methadone | Buprenorphine/Naloxone | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 25 | 53
  >=65 years | 0 | 1 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 37.7 (8.6) | 39.0 (10.9) | 38.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 25
  Male | 12 | 17 | 29
Region of Enrollment [Number; unit: participants]
  United States | 28 | 26 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Retained in Treatment
Description: This outcome assesses the number of participants who completed the treatment after 6 months.
Time Frame: 6 months
Population: All participants that were randomized were analyzed regarding their retention in treatment at 6 months.
Measure: Number; unit: participants
Groups:
- Methadone: Methadone 10-60 mg per day divided in 2-4 doses for 6 months
- Buprenorphine/Naloxone: Buprenorphine 4-16 mg per day divided in 2-4 doses for 6 months (using tablets of buprenorphine/naloxone:4/1 mg)
Arm/Group | Methadone | Buprenorphine/Naloxone
Number analyzed (Participants) | 28 | 26
participants | 13 | 13
Statistical Analysis 1: Comparison: Methadone vs Buprenorphine/Naloxone; Null hypothesis: Methadone and buprenorphine treatment do not differ in treatment retention; Test type: Superiority or Other; p = 0.77, Log Rank; Hazard Ratio (HR) = 0.9134, 95% CI 2-sided [0.4156 to 2.007]

2. Secondary Outcome: Numerical Rating Score for Pain
Description: Pain was measured using a 0-10 point numerical rating scale (NRS) with 0 representing no pain and 10 representing worst pain possible.
Time Frame: 6 months
Population: Participants that completed the treatment at 6 months were analyzed.
Measure: Mean (Standard Deviation); unit: units on a 0-10 NRS scale
Arm/Group | Methadone | Buprenorphine/Naloxone
Number analyzed (Participants) | 13 | 13
units on a 0-10 NRS scale | 5.4 (1.1) | 5.6 (2.5)
Statistical Analysis 1: Comparison: Methadone vs Buprenorphine/Naloxone; Null hypothesis: Methadone treatment is as effective as buprenorphine treatment in reducing pain; Test type: Superiority or Other; p < 0.043, ANOVA; Mean Difference (Final Values) = 0.2

3. Secondary Outcome: Numerical Rating Score for Functioning
Description: We assessed functioning measured on a 0-10 point numerical rating scale (NRS)with 0 being the least amount of functioning and 10 the best amount of functioning.
Time Frame: 6 months
Population: The participants who completed the treatment were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: units on a 0-10 point NRS scale
Arm/Group | Methadone | Buprenorphine/Naloxone
Number analyzed (Participants) | 13 | 13
units on a 0-10 point NRS scale | 5.0 (1.7) | 5.3 (2.0)
Statistical Analysis 1: Comparison: Methadone vs Buprenorphine/Naloxone; null-hypothesis: methadone and buprenorphine treatment are equally effective in reducing self-reported functioning at 6 months; Test type: Superiority or Other; p < 0.665, ANOVA; Mean Difference (Final Values) = 0.3, Standard Deviation 0

4. Secondary Outcome: Self-reported Illicit Opioid Use
Time Frame: 6 months
Measure: Number; unit: number of participants
Arm/Group | Methadone | Buprenorphine/Naloxone
Number analyzed (Participants) | 13 | 13
number of participants | 0 | 5
Statistical Analysis 1: Comparison: Methadone vs Buprenorphine/Naloxone; Null hypothesis: methadone or buprenorphine treatment equally reduce illicit drug use; Test type: Superiority or Other; p < 0.039, Fisher Exact; Odds Ratio (OR) = 0, Standard Deviation 0

ADVERSE EVENTS:
Arm/Group | Methadone | Buprenorphine/Naloxone
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/26
Other Adverse Events (participants affected / at risk) | 0/28 | 0/26

LIMITATIONS AND CAVEATS:
small subject number not a double-blind study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No